CLINICAL TRIAL: NCT02810223
Title: Efficacy of CART-19 Cell Therapy in B Cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sanwater Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT1601-CART19
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-06

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose of CART-19 (Experimental): 2 to 5 x 10(6) autologous CART-19 transduced cells per kg body weight, with a maximum dose of 2.5 x 10(8) autologous CTL019 transduced cells via intravenous infusion.
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — 2 to 5 x 10(6) autologous CART-19 transduced cells per kg body weight, with a maximum dose of 2.5 x 10(8) autologous CTL019 transduced cells via intravenous infusion.

SUMMARY:
This is a single arm, open-label, multi-center study to determine the efficacy and safety of an experimental therapy called CART-19 in patients with chemo-refractory and relapsed B-cell ALL.

DETAILED DESCRIPTION:
This is a single arm, open-label, multi-center, phase I study to determine the efficacy of CTL019 in patients with r/r B-cell ALL. The study will have the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Primary Follow-up, Secondary Follow-up (if applicable) and Survival Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD 19+ B cell acute lymphoblastic leukemia in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to <2 year survival) with currently available therapies will be enrolled

  1. Age 1 to 60 years.
  2. Expected survival > 12 weeks
  3. Creatinine < 2.5 mg/dl and less than 2.5x normal for age
  4. ALT ≤ 5x normal
  5. Bilirubin <2.0 mg/dl
  6. Any relapse after prior SCT will make patient eligible regardless of other prior therapy
  7. Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and

     ①. Have no active GVHD and require no immunosuppression

     ②. Are more than 4 months from transplant
  8. For those patients who require leukapheresis for T cell collection (i.e. no previously collected product exists), adequate venous access for apheresis or eligible for appropriate catheter placement, and no other contraindications for leukapheresis
  9. Voluntary informed consent is given
  10. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy (at infusion)

      Exclusion Criteria:

  <!-- -->

  1. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
  2. Uncontrolled active infection
  3. Active hepatitis B or hepatitis C infection
  4. Concurrent use of systemic steroids at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of inhaled steroids, or hydrocortisone for physiological replacement in patients with adrenal insufficiency are permitted as well
  5. Presence of grade 2-4 acute or extensive chronic GVHD
  6. Under treatment for GVHD
  7. Previous treatment with any gene therapy products
  8. Any uncontrolled active medical disorder that would preclude participation as outlined.
  9. HIV infection.
  10. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided